CLINICAL TRIAL: NCT02180737
Title: Evaluation of Role of Dexmedetomidine as a Sole Agent in Sedation of Cancer Patients Undergoing Radiological Interventional Procedures
Brief Title: Dexmedetomidine for Sedation During Radiological Interventional Procedures
Acronym: Dexmed
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ghada M N Bashandy, Dr, National Cancer Institute, Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dexmedetomidine sedation
Record Dates: First submitted 2014-06-30; First posted 2014-07-03 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Procedural Sedation
Keywords: dexmedetomedine; sedation; interventional radiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dexmeditomedine (Experimental): Dexmedetomidine will be initiated at 0.6 mcg/kg/hr and titrated to achieve desired clinical effect with doses ranging from 0.2 to 1 mcg/kg/hr.
  Interventions: Drug: Dexmeditomedine

INTERVENTIONS:
Drug: Dexmeditomedine
  Other Names: Dexmedetomidine at 0.6 mcg/kg/hr then 0.2 to 1 mcg/kg/hr.

SUMMARY:
Evaluation of the role of dexmedetomidine as a sole agent in sedating patients undergoing interventional radiological procedures and measuring its different outcome variables.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18-65 years old
* ASA physical status of I-II
* Expected procedure lasting at least 30 minutes

Exclusion Criteria:

* Unstable cardiac status (life-threatening arrhythmias, abnormal cardiac anatomy, significant cardiac dysfunction and third-degree heart block.
* An alpha2-agonist or antagonist within 14 days before the scheduled procedure.
* patients received an IV opioid within 1 h, or an oral or IM opioid within 4 h of the start of study drug administration.
* Patients who are allergic to Dexmedetomidine or alpha 2-agonists.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Degree of sedation | 1 hour
  It will be measured and recorded by using the Ramsay sedation score.
verbal analogue scale | 1 hour
  assessment of pain using VAS score

SECONDARY OUTCOMES:
patient satisfaction | 24 hours
  assessment of patient satisfaction by 4 point scale

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa T Salem, MD, Study Chair — National Cancer Institute (NCI); Maie K Helaly, MD, Study Director — National Cancer Institute (NCI); Ghada M Bashandy, MD, Principal Investigator — National Cancer Institute (NCI); Ayat A Hassan, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute-Egypt, Cairo, Egypt

REFERENCES:
- [Result] Hsu YW, Cortinez LI, Robertson KM, Keifer JC, Sum-Ping ST, Moretti EW, Young CC, Wright DR, Macleod DB, Somma J. Dexmedetomidine pharmacodynamics: part I: crossover comparison of the respiratory effects of dexmedetomidine and remifentanil in healthy volunteers. Anesthesiology. 2004 Nov;101(5):1066-76. doi: 10.1097/00000542-200411000-00005. PMID 15505441
- [Result] Scher CS, Gitlin MC. Dexmedetomidine and low-dose ketamine provide adequate sedation for awake fibreoptic intubation. Can J Anaesth. 2003 Jun-Jul;50(6):607-10. doi: 10.1007/BF03018650. PMID 12826556